CLINICAL TRIAL: NCT03500276
Title: Impact of Yoga on Quality of Life and Markers of Inflammation in Rheumatoid Arthritis Patients
Brief Title: Yoga for Patients With Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Dubrava (Other)
Responsible Party: Principal Investigator, SILVA PUKŠIĆ, MD, PhD candidate, University Hospital Dubrava
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DUBRAVA-YOGRA-01
Record Dates: First submitted 2018-04-07; First posted 2018-04-18 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Rheumatoid Arthritis
Keywords: yoga; health-related quality of life; proinflammatory genes; inflammatory markers; rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial
Who Masked: Outcomes Assessor
Masking Description: Blinded rater will be used to assess disease activity by DAS28CRP score.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga program (Experimental): 12 weeks of "Yoga in daily life practice", 2x weekly for 90 minutes including physical exercises (asanas), breathing exercises (pranayama), relaxation and meditation exercises.
  Interventions: Behavioral: Yoga program
- Arthritis-education control (Active Comparator): 12 weeks of arthritis - education classes, consisting of 1x weekly sessions for 120 minutes including lectures on arthritis and related issues followed by group discussion.
  Interventions: Behavioral: Arthritis-education

INTERVENTIONS:
Behavioral: Yoga program — Yoga classes will be conducted 2xweekly/ 90 minutes and consist of physical exercises (asanas), breathing exercises (pranayama), relaxation and self-enquiry meditation based on Yoga in daily life system.
  Arms: Yoga program
Behavioral: Arthritis-education — Arthritis-education classes will be conducted 1xweekly/ 120 minutes and led by rheumatology specialists and consist of lectures on arthritis and related issues followed by group discussion.
  Arms: Arthritis-education control

SUMMARY:
The purpose of this study is to investigate the effects of a yoga program based on "Yoga in daily life system" in patients with rheumatoid arthritis.

The investigators want to explore whether this program will improve health-related quality of life and psychological well-being in patients. In addition they want to explore its potential positive modulation of the immune system.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic disabling inflammatory disease that substantially impacts health-related quality of life (HRQOL) of patients. In addition to pain, fatigue and physical disability the disease also affects psychological health. Yoga, a mind-body therapy, integrates physical exercises with relaxation and meditation. Published data suggest its beneficial effects on both physical and mental health in various chronic conditions. The true biological mechanism underlying these effects is not well known. Recent research suggests potential modulation of the immune system and inflammation-related gene expression changes.

Hypothesis: Yoga program based on Yoga in daily life system has positive impact on clinical and biologic outcomes in RA patients.

Aims: To determine the impact of a 12-week yoga program on measures of psychological distress, HRQOL, fatigue, pain, disease activity, levels of circulating inflammatory markers and pro-inflammatory gene expression.

Materials and methods: 50 RA patients, aged 18-65 years, on stable standard pharmacological treatment will be randomly assigned to a 12-week yoga intervention (based on "Yoga in daily life system") or arthritis-education control. Self-administered questionnaires will be used to assess quality of life and psychological well-being of the patients. Blood samples will be collected for measurement of inflammatory markers and expression of a set of pro-inflammatory genes. Disease activity will be assessed by DAS28CRP score. The patients will be assessed on baseline, post-treatment and at 3 months follow-up.

This research will provide information on potential efficacy of yoga program in improving physical and psychological outcomes in persons with RA and explore its influence on immunological system.

ELIGIBILITY:
Inclusion Criteria:

1. ACR/EULAR 2010. classification criteria for rheumatoid arthritis (RA)
2. disease activity measured by DAS28CRP< 5.1
3. patients on stable dose of disease-modifying antirheumatic medications,non-steroidal anti-inflammatory drugs or low-dose glucocorticoids for the last 3 months

Exclusion Criteria:

1. significant co-morbidity (active malignant disease, symptomatic ischemic heart disease or heart failure, severe lung disease, uncontrolled thyroid disease, neurological disease that impairs mobility) that is more limiting than RA
2. history of drug or alcohol abuse
3. recent injury/ or surgery
4. regular practice of yoga or similar technique in the last 6 months or currently engaged in a structured exercise program for >=2 times weekly, patients that are currently engaged in physical therapy
5. pregnant or planning pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Change in health-related quality of life | baseline and 12 weeks
  The Medical Outcomes Survey 36-item Short-Form Healthy Survey ( SF-36). A 36 item generic health survey measures general health concepts through 8 domains: physical functioning, role physical, bodily pain, global health, vitality, social functioning, role emotional, mental health. Scores 0-100, with higher scores indicating better health

SECONDARY OUTCOMES:
Change in pro-inflammatory gene expression | baseline and 12 weeks
  RT-PCR analysis of expression of a set of pro-inflammatory genes. Changes from baseline to 12 weeks
Change in blood levels of hs-CRP | baseline and 12 weeks
  hs-CRP (mg/l) changes from baseline to 12 weeks
Change in blood levels of hs-CRP | baseline and 24 weeks
  hs-CRP (mg/l) changes from baseline to 24 weeks
Change in pain intensity | baseline and 12 weeks
  Visual analogue scale 0-10, with higher scores indicating higher pain intensity
Change in pain intensity | baseline and 24 weeks
  Visual analogue scale 0-10, with higher scores indicating higher pain intensity
Change in perceived stress | baseline and 12 weeks
  Perceived Stress Scale (PSS) consists of 10 items. Range 0-40 points with higher scores indicating greater levels of stress
Change in perceived stress | baseline and 24 weeks
  Perceived Stress Scale (PSS) consists of 10 items. Range 0-40 points with higher scores indicating greater levels of stress
Change in rheumatoid arthritis activity | baseline and 12 weeks
  Disease Activity Score 28 (DAS28CRP). Composite index including a non-graded 28 tender and swollen joint count, patients global health (VAS-GH scored 0-100), and CRP in mg/l. It is based on a complex equasion DAS28 = 0.56 × √[t28] + 0.28 × √[sw28] + 0.70 × Ln [CRP] + 0.014 × GH. Lower range 0, no higher range. Higher levels indicating higher disease activity
Change in rheumatoid arthritis activity | baseline and 24 weeks
  Disease Activity Score 28 (DAS28CRP). Composite index including a non-graded 28 tender and swollen joint count, patients global health (VAS-GH scored 0-100), and CRP in mg/l. It is based on a complex equasion DAS28 = 0.56 × √[t28] + 0.28 × √[sw28] + 0.70 × Ln [CRP] + 0.014 × GH. Lower range 0, no higher range. Higher levels indicating higher disease activity
Change in fatigue intensity | baseline and 12 weeks
  Functional assessment of chronic illness therapy - fatigue (FACIT-F) scale consisting of 13 items. Range 0-52 with higher scores indicating higher levels of fatigue
Change in fatigue intensity | baseline and 24 weeks
  Functional assessment of chronic illness therapy - fatigue (FACIT-F) scale consisting of 13 items. Range 0-52 with higher scores indicating higher levels of fatigue
Change in anxiety and depression symptoms | baseline and 12 weeks
  Hospital anxiety and depression scale (HADS) measures levels of anxiety and depression (total score range 0-42 points) consists of subscale for anxiety 0-21 points and sub-scale for depression 0-21 points. Higher scores indicate higher levels of anxiety / depression.
Change in anxiety and depression symptoms | baseline and 24 weeks
  Hospital anxiety and depression scale (HADS) measures levels of anxiety and depression (total score range 0-42 points) consists of subscale for anxiety 0-21 points and sub-scale for depression 0-21 points. Higher scores indicate higher levels of anxiety / depression.
Change in rheumatoid arthritis impact of disease | baseline and 12 weeks
  Rheumatoid arthritis impact of disease questionnaire (RAID) is a patient-derived scores assessing 7 most important domains of impact of rheumatoid arthritis. Domains include pain, functional disability, fatigue, emotional and physical well-being, sleep and coping. Range 0-10.Higher scores reflect higher levels of symptoms.
Change in rheumatoid arthritis impact of disease | baseline and 24 weeks
  Rheumatoid arthritis impact of disease questionnaire (RAID) is a patient-derived scores assessing 7 most important domains of impact of rheumatoid arthritis. Domains include pain, functional disability, fatigue, emotional and physical well-being, sleep and coping. Range 0-10.Higher scores reflect higher levels of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Silva Pukšić, MD, Principal Investigator — University Hospital Dubrava; Jadranka Morović-Vergles, MD, PhD, Study Chair — University Hospital Dubrava
Locations (1):
- University Hospital Dubrava, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No